CLINICAL TRIAL: NCT02319642
Title: A Phase 3, Multicenter, Open-label Extension Study To Assess The Safety And Efficacy Of Certolizumab Pegol As Additional Medication To Methotrexate In Chinese Subjects With Active Rheumatoid Arthritis Who Participated In RA0044.
Brief Title: An Open-label Extension Study of Certolizumab Pegol in Chinese Patients With Rheumatoid Arthritis Who Enrolled in RA0044
Acronym: RAPID-C OLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA0078; CTR20140412 (Other: www.ChinaDrugTrials.org)
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; TNFα antagonist; Certolizumab pegol; Chinese patients; Open-label
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Certolizumab Pegol (CZP) (Experimental): 1. Those subjects from either treatment group in RA0044 (NCT02151851) who fail to achieve an ACR20 response in RA0044 (NCT02151851) at Week 12, which is confirmed at Week 14. These subjects are withdrawn from RA0044 (NCT02151851) at Week 16 of that study, and that assessment will also be the Entry assessment for this Extension study. In this OLE study, these subjects will receive CZP 400 mg sc at Weeks 0, 2, and 4 followed by CZP 200 mg sc Q2W.
  2. Subjects from either treatment group in RA0044 (NCT02151851) who completed RA0044 (NCT02151851) through Week 24. The Week 24 assessment in RA0044 (NCT02151851) will also be the Entry assessment for this Extension study. In this OLE study, these subjects will receive CZP 200 mg sc Q2W.
  Interventions: Drug: Certolizumab Pegol

INTERVENTIONS:
Drug: Certolizumab Pegol — Active Substance: Certolizumab Pegol Pharmaceutical form: Prefilled syringes Concentration: 200 mg/ ml Route of Administration: Subcutaneous injection
  Other Names: Cimzia

SUMMARY:
This study will continue to evaluate the safety & efficacy of Certolizumab Pegol (CZP) for 6 months in Chinese subjects with active Rheumatoid Arthritis who participated in RA0044.

DETAILED DESCRIPTION:
This study (RA0078) will continue to assess the safety, tolerability, and efficacy of Certolizumab Pegol (CZP) for 6 months as additional medication to methotrexate (MTX) with or without folic acid in Chinese subjects with active Rheumatoid Arthritis (RA) who participated in the main feeder study, RA0044. All subjects will continue to receive their established treatment with MTX with or without folic acid. The dose of MTX may be decreased by the Investigator due to toxicity, but should not be discontinued completely. Concomitant nonsteroidal anti-inflammatory drugs and oral corticosteroids will be permitted. For each subject, the study duration will last a maximum of approximately 32 weeks.

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board (IRB)/ Independent Ethics Committee (IEC) approved written Informed Consent form (ICF) for RA0078 is signed and dated by the subject or by the parent(s) or legal representative
* Subject/ legal representative is considered reliable and capable of adhering to the protocol (eg, able to understand and complete diaries), visit schedule, and medication intake according to the judgment of the Investigator
* Subjects must either have:

  * Completed RA0044 through Week 24, OR
  * Failed to achieve an ACR20 response at Week 12 (confirmed at Week 14) in RA0044
* Subjects must have complied with the protocol requirements during their participation in RA0044
* Subjects entering RA0078 who have completed RA0044 must have a clear chest x-ray at the Week 24 Completion Visit of RA0044. Subjects who enter RA0078 at Week 16 of the RA0044 study are not required to have a chest x-ray prior to enrollment
* Subject is able to continue treatment with Methotrexate (MTX) (with or without folic acid) at a dose deemed appropriate by the Investigator
* Female subjects with childbearing potential should have a negative pregnancy test at Entry and should have a medically accepted method of contraception used during the entire duration of the study and for 10 weeks after the last dose of Certolizumab pegol (CZP). Medically accepted methods of contraception are: hormonal contraception for at least 2 cycles prior to Screening, intrauterine device, implant device, diaphragm with spermicide, bilateral tubal ligation, monogamous relationship with vasectomized (for at least 3 months prior to Screening) partner, or using condoms with spermicide gel. Abstinence is not an acceptable method of contraception for the study. Female subjects who are postmenopause for at least 2 years or had undergone a complete hysterectomy, bilateral tubal ligation and/ or bilateral ovariectomy, or have a congenital sterility are considered not of childbearing potential. Male subjects must agree to ensure they use adequate contraception during the study and for at least 10 weeks after the subject receives their last dose of study medication

Exclusion Criteria:

Rheumatoid Arthritis (RA) disease-related exclusions:

* Subjects have a diagnosis of any other inflammatory arthritis eg, psoriatic arthritis or ankylosing spondylitis
* Subjects have a secondary, noninflammatory type of arthritis (eg, osteoarthritis or fibromyalgia) that in the Investigator's opinion is symptomatic enough to interfere with evaluation of the effect of CZP on the subject's primary diagnosis of RA
* Subjects have a history of an infected joint prosthesis at any time with that prosthesis still in situ

Concomitant medication exclusions

* Subjects must be free of the following concomitant medications:

  * Any biological therapy for RA
  * Any experimental therapy, within or outside a clinical trial (except RA0044)
  * Live vaccines Medical history exclusions
* Lactating and/or pregnant female subjects
* Male subjects with childbearing potential partner(s) and female subjects of childbearing potential who are NOT practicing effective birth control. All female subjects must test negative on a urine pregnancy test before study entry and at each study visit
* Subjects with known TB infection, at high risk of acquiring TB infection, or latent TB (LTB) infection (with exception) are excluded
* Subjects who had 3 or more infections requiring systemic antibiotics during RA0044
* Subjects with a history of chronic infection, recent serious or life-threatening infection (within 6 months, including herpes zoster), or a current sign or symptom that may indicate an infection (eg, fever, cough)
* Subjects with a history or active systemic/ respiratory infection due to fungal, parasitic, or mycotic pathogens including but not limited to histoplasmosis, coccidiosis, paracoccidiosis, pneumocystis, blastomyces, aspergillus, and nontuberculous mycobacteria (NTMB)
* Radiographic evidence suggestive of any of these infections is sufficient grounds for exclusion
* Subjects at a high risk of infection in the Investigator's opinion (eg, subjects with leg ulcers, indwelling urinary catheter, and persistent or recurrent chest infections, and subjects who are permanently bedridden or wheelchair bound)
* Subjects with a known positive hepatitis B surface antigen (HBsAg) test and/ or hepatitis C virus antibody (anti-HCV) test result
* Subjects with known human immunodeficiency virus (HIV) infection
* Subjects with lymphoproliferative disorder including lymphoma or signs and symptoms suggestive of lymphoproliferative disease at any time
* Subjects with active malignancy of any type
* Subjects with a history of blood dyscrasias, eg, leukemia or hemophilia where the blood constituents are abnormal or are present in abnormal quantity.
* Subjects with class III or IV congestive heart failure New York Heart Association (NYHA) 1994
* Subjects with suspected or diagnosed demyelinating disease of the central nervous system (eg, multiple sclerosis or optic neuritis)
* Subjects with a current or recent history, as determined by the Investigator, of severe, progressive, and/or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, or cerebral disease which would interfere with the subject's participation in the study. Abnormal laboratory parameters that require exclusion of a subject are detailed in protocol
* Subjects with an adverse reaction to Percutaneous Endoscopic Gastrostomy (PEG) or a protein medicinal product or known hypersensitivity to any components of the study medication or comparative drugs as stated in this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2014-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 887.822.9493
Locations (30):
- China (30):
  - 037, Baotou
  - 001, Beijing
  - 002, Beijing
  - 013, Beijing
  - 021, Beijing
  - 025, Beijing
  - 033, Beijing
  - 014, Bengbu
  - 034, Changchun
  - 017, Changsha
  - 019, Changsha
  - 007, Chengdu
  - 012, Chengdu
  - 004, Guangzhou
  - 015, Hangzhou
  - 005, Hefei
  - 008, Heilongjiang
  - 011, Jilin
  - 022, Jinan
  - 031, Kunming
  - 028, Nanjing
  - 009, Shanghai
  - 018, Shanghai
  - 020, Shanghai
  - 030, Shanghai
  - 038, Shijiazhuang
  - 010, Tianjin
  - 006, Wuhan
  - 016, Xi'an
  - 035, Xi'an

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll subjects in November 2014 and concluded in December 2016.
Pre-assignment Details: Participant Flow refers to the Safety Set consisting of all subjects who were dispensed medication.
Groups:
- Open-label Cimzia (Placebo in Feeder Study): Subjects were treated with Placebo in the feeder study RA0044 (NCT02151851). In this OLE study, these subjects received either CZP 400 mg subcutaneously (sc) at Weeks 0, 2, and 4 followed by CZP 200 mg sc every two weeks (Q2W) if they fail to achieve an ACR20 response in RA0044 (NCT02151851) at Week 12, which is confirmed at Week 14 or CZP 200 mg sc Q2W if they completed RA0044 (NCT02151851) through week 24.
- Open-label Cimzia (Cimzia in Feeder Study): Subjects were treated with CZP in the feeder study RA0044 (NCT02151851). In this OLE study, these subjects receive either CZP 400 mg sc at Weeks 0, 2, and 4 followed by CZP 200 mg sc Q2W if they fail to achieve an ACR20 response in RA0044 (NCT02151851) at Week 12, which is confirmed at Week 14 or CZP 200 mg sc Q2W if they completed RA0044 (NCT02151851) through week 24.
Period: Overall Study
Arm/Group | Open-label Cimzia (Placebo in Feeder Study) | Open-label Cimzia (Cimzia in Feeder Study)
Started | 95 | 251
Completed | 91 | 245
Not Completed | 4 | 6
Not completed — Adverse Event | 2 | 4
Not completed — Lack of Efficacy | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set. Demographic baseline refers to RA0044 (NCT02151851) baseline with a subset of subjects who enrolled into RA0078.
Arm/Group | Open-label Cimzia (Placebo in Feeder Study) | Open-label Cimzia (Cimzia in Feeder Study) | Total Title
Number analyzed (Participants) | 95 | 251 | 346
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 91 | 239 | 330
  >=65 years | 4 | 12 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (10.9) | 47.5 (11.6) | 47.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 216 | 293
  Male | 18 | 35 | 53

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects That Withdrew Due to a Treatment-emergent Adverse Event (TEAE)
Description: TEAEs are defined as Advere Events (AEs) starting on or after the date of first study medication administration in this Open-label Extension (OLE) study up to 70 days post-last dose.
Time Frame: Baseline to the end of observation period (32 weeks)
Population: Safety Set
Measure: Number; unit: percentage of participants
Arm/Group | Open-label Cimzia (Placebo in Feeder Study) | Open-label Cimzia (Cimzia in Feeder Study)
Number analyzed (Participants) | 95 | 251
percentage of participants | 2.1 | 1.6

2. Primary Outcome: Percentage of Subjects With at Least One Treatment-emergent Adverse Event (TEAE)
Description: TEAEs are defined as Adverse Events (AEs) starting on or after the date of first study medication administration in this Open-label Extension (OLE) study up to 70 days post-last dose.
Time Frame: Baseline to the end of observation period (32 weeks)
Population: Safety Set
Measure: Number; unit: percentage of participants
Groups:
- Open-label Cimzia (Placebo in Feeder Study): Subjects were treated with Placebo in study RA0044 (NCT02151851). In this OLE study, these subjects received either CZP 400 mg subcutaneously (sc) at Weeks 0, 2, and 4 followed by CZP 200 mg sc every two weeks (Q2W) if they fail to achieve an ACR20 response in RA0044 (NCT02151851) at Week 12, which is confirmed at Week 14 or CZP 200 mg sc Q2W if they completed RA0044 (NCT02151851) through week 24.
- Open-label Cimzia (Cimzia in Feeder Study): Subjects were treated with CZP in study RA0044 (NCT02151851). In this OLE study, these subjects receive either CZP 400 mg sc at Weeks 0, 2, and 4 followed by CZP 200 mg sc Q2W if they fail to achieve an ACR20 response in RA0044 (NCT02151851) at Week 12, which is confirmed at Week 14 or CZP 200 mg sc Q2W if they completed RA0044 (NCT02151851) through week 24.
Arm/Group | Open-label Cimzia (Placebo in Feeder Study) | Open-label Cimzia (Cimzia in Feeder Study)
Number analyzed (Participants) | 95 | 251
percentage of participants | 65.3 | 65.3

3. Primary Outcome: Percentage of Subjects With at Least One Treatment-emergent Serious Adverse Event (SAE)
Description: Treatment emergent SAEs are defined as SAEs starting on or after the date of first study medication administration in this OLE study up to 70 days post-last dose.
Time Frame: Baseline to the end of observation period (32 weeks)
Population: Safety Set
Measure: Number; unit: percentage of participants
Arm/Group | Open-label Cimzia (Placebo in Feeder Study) | Open-label Cimzia (Cimzia in Feeder Study)
Number analyzed (Participants) | 95 | 251
percentage of participants | 6.3 | 2.0

4. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20 (ACR20) in Relation to Baseline
Description: The ACR20 represents improvement from Baseline of at least 20 %, calculated from assessments of tender joint count, swollen joint count, Patient's Assessment of Arthritis Pain (PtAAP) -visual analog scale (VAS), Patient's Global Assessment of Disease Activity (PtGADA) -VAS, Physician's Global Assessment of Disease Activity (PhGADA) -VAS, Health Assessment Questionnaire-Disability Index (HAQ-DI), and C-reactive protein (CRP).
  Responder was relative to baseline of RA0044. Baseline value in RA0044 was defined as the last non-missing measurement collected prior to first study drug administration in RA0044.
Time Frame: Week 24
Population: Safety Set with Non-Responder-Imputation (NRI).
Measure: Number; unit: percentage of participants
Arm/Group | Open-label Cimzia (Placebo in Feeder Study) | Open-label Cimzia (Cimzia in Feeder Study)
Number analyzed (Participants) | 95 | 251
percentage of participants | 72.6 | 82.1

5. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 50 (ACR50) in Relation to Baseline
Description: The ACR50 represents improvement from Baseline of at least 50 %, calculated from assessments of tender joint count, swollen joint count, Patient's Assessment of Arthritis Pain (PtAAP) -visual analog scale (VAS), Patient's Global Assessment of Disease Activity (PtGADA) -VAS, Physician's Global Assessment of Disease Activity (PhGADA) -VAS, Health Assessment Questionnaire-Disability Index (HAQ-DI), and C-reactive protein (CRP).
  Responder was relative to baseline of RA0044. Baseline value in RA0044 was defined as the last non-missing measurement collected prior to first study administration in RA0044.
Time Frame: Week 24
Population: Safety Set with Non-Responder-Imputation (NRI).
Measure: Number; unit: percentage of participants
Arm/Group | Open-label Cimzia (Placebo in Feeder Study) | Open-label Cimzia (Cimzia in Feeder Study)
Number analyzed (Participants) | 95 | 251
percentage of participants | 45.3 | 56.6

6. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 70 (ACR70) in Relation to Baseline
Description: The ACR70 represents improvement from Baseline of at least 70 %, calculated from assessments of tender joint count, swollen joint count, Patient's Assessment of Arthritis Pain (PtAAP) -visual analog scale (VAS), Patient's Global Assessment of Disease Activity (PtGADA) -VAS, Physician's Global Assessment of Disease Activity (PhGADA) -VAS, Health Assessment Questionnaire-Disability Index (HAQ-DI), and C-reactive protein (CRP).
  Responder was relative to baseline of RA0044. Baseline value in RA0044 was defined as the last non-missing measurement collected prior to first study administration in RA0044.
Time Frame: Week 24
Population: Safety Set with Non-Responder-Imputation (NRI).
Measure: Number; unit: percentage of participants
Arm/Group | Open-label Cimzia (Placebo in Feeder Study) | Open-label Cimzia (Cimzia in Feeder Study)
Number analyzed (Participants) | 95 | 251
percentage of participants | 17.9 | 31.5

7. Secondary Outcome: Change From Baseline Value in Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: Each subject will complete the HAQ-DI questionnaire at the visit and provides an assessment of the impact of the disease and its treatment on physical function. HAQ-DI scores range from 0 to 3. Lower scores indicate less disability.
  Negative values indicate improvement from Baseline. Baseline refers to RA0044 baseline.
Time Frame: Week 24
Population: Safety Set with last observation carried forward (LOCF). Only subjects with available data are included in the analysis of this Outcome Measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Cimzia (Placebo in Feeder Study) | Open-label Cimzia (Cimzia in Feeder Study)
Number analyzed (Participants) | 95 | 251
units on a scale | -0.526 (0.621) | -0.681 (0.611)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Baseline of RA0078 until Safety Follow Up visit (up to Week 32).
Description: Adverse Events refer to the Safety Population consisting of all subjects who were dispensed medication.
Arm/Group | Open-label Cimzia (Placebo in Feeder Study) | Open-label Cimzia (Cimzia in Feeder Study)
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/251
Serious Adverse Events (participants affected / at risk) | 6/95 | 5/251
Other Adverse Events (participants affected / at risk) | 21/95 | 55/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Cimzia (Placebo in Feeder Study) (N=95) | Open-label Cimzia (Cimzia in Feeder Study) (N=251)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Cimzia (Placebo in Feeder Study) (N=95) | Open-label Cimzia (Cimzia in Feeder Study) (N=251)
Anaemia (Blood and lymphatic system disorders) | 5 (7) | 14 (15)
Upper respiratory tract infection (Infections and infestations) | 13 (14) | 39 (45)
Liver function test abnormal (Investigations) | 5 (8) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days